CLINICAL TRIAL: NCT03928223
Title: The Color of Itch; Itch Modification by Color Viewing- an Exploratory Survey
Brief Title: The Color of Itch; Itch Modification by Color Viewing
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req 2017-1; sp19Mueller4
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Itch; Pruritus
Keywords: contagious itch; Manchester Color Wheel
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exploratory survey on Itch modification by color viewing — Patients relate their itch to a color of the Manchester Color Wheel (MCW) and choose a color of the MCW aimed at counteracting their itch. They complete the ItchyQoL (German version), which is a standard tool to assess itch-related quality of life. Then patients look at their "antipruritic" monochrome color for five minutes on a lap-top screen. Itch intensity (0-10 NRS) will be assessed at baseline and again after the patients looked at this color for 5 minutes.

SUMMARY:
Itch is the commonest skin-related symptom. There is increasing evidence that itch can be influenced by visual cues. The impact of colors on itch has not yet been studied.

This study investigates Itch modification by color viewing and whether patients can match or counteract their itch with a color.

ELIGIBILITY:
Inclusion Criteria:

* Dermatology in- and outpatients with itch

Exclusion Criteria:

* color blindness
* lack of time
* lack of German language.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dermatology in- and outpatients with itch in the Department of Dermatology of the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in itch intensity | assessed at baseline and again after the patients looked at the "antipruritic" color for 5 minutes
  Change in itch intensity (measured on a 0-10 Numerical Rating Scale, NRS); 0 = no itch; 10 = most intensive itch

CONTACTS AND LOCATIONS:
Overall Officials: Simon Müller, Dr. med, Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland